CLINICAL TRIAL: NCT02807350
Title: A Randomized Clinical Trial of Overminus Spectacle Therapy for Intermittent Exotropia
Brief Title: Trial of Overminus Spectacle Therapy for Intermittent Exotropia
Acronym: IXT5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IXT5; 2U10EY011751 (NIH)
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Results first posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Intermittent Exotropia
Keywords: Intermittent Exotropia; IXT; overminus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Overminus Treatment (Experimental): spectacles with full cycloplegic refraction plus 2.50 D overminus added to the sphere
  Interventions: Device: Overminus treatment
- Non-overminus Treatment (Active Comparator): spectacles with full cycloplegic refraction without overminus
  Interventions: Device: Non-overminus treatment

INTERVENTIONS:
Device: Overminus treatment — spectacles with full cycloplegic refraction plus 2.50 D overminus added to the sphere
  Other Names: Overminus spectacles; Overminus glasses; Overminus therapy
  Arms: Overminus Treatment
Device: Non-overminus treatment — spectacles with full cycloplegic refraction without overminus
  Arms: Non-overminus Treatment

SUMMARY:
The main objectives of this randomized trial comparing overminus lens treatment to non-overminus (spectacles without overminus or spectacles with plano lenses) are to determine:

* The long-term on-treatment effect of overminus treatment on distance intermittent exotropia (IXT) control score.
* The off-treatment effect of overminus treatment on distance IXT control score (following weaning and 3 months off treatment).

DETAILED DESCRIPTION:
The main objectives of this randomized trial comparing overminus lens treatment to non-overminus (spectacles without overminus or spectacles with plano lenses) are to determine:

* The long-term on-treatment effect of overminus treatment on distance IXT control score.
* The off-treatment effect of overminus treatment on distance IXT control score (following weaning and 3 months off treatment).

The recently completed IXT3 pilot study (NCT02223650) addressed the question of whether overminus lens therapy has an initial short-term therapeutic effect for IXT while wearing overminus spectacles. There have been no rigorous studies that address the following important questions related to overminus lens therapy:

* Does overminus lens therapy have a long-term therapeutic effect for IXT while wearing overminus spectacles (over many months or years)?
* Does overminus lens therapy have a long-term therapeutic effect for IXT when overminus spectacles are discontinued?

In November 2019, a protocol amendment discontinued overminus lens treatment and extended the study for an additional 18 months after the 18-month randomized trial has ended. The objective of the extension study is to compare long-term refractive error between subjects originally treated with either overminus spectacles or non-overminus spectacles as part of the 18-month randomized trial; treatment is at investigator discretion.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 years to < 11 years
* Intermittent exotropia (manifest deviation) meeting all of the following criteria:
* At distance: intermittent exotropia or constant exotropia

  o Mean distance control score of 2 points or more (mean of 3 assessments over the exam)
* At near: intermittent exotropia, exophoria, or orthophoria

  o Subject cannot have a score of 5 points on all 3 near assessments of control
* Exodeviation at least 15∆ at distance measured by PACT
* Near deviation does not exceed distance deviation by more than 10∆ by PACT (convergence insufficiency type IXT excluded)
* Distance visual acuity (any optotype method) in each eye of 0.4 logMAR (20/50) or better if age 3 years and 0.3 logMAR (20/40) or better if 4 years or older.
* Interocular difference of distance visual acuity ≤0.2 logMAR (2 lines on a logMAR chart)
* Refractive error between -6.00 diopters (D) standard error (SE) and +1.00D SE (inclusive) in the most myopic / least hyperopic eye based on a cycloplegic refraction performed within the past 2 months or at the end of the enrollment exam.
* If refractive error (based on cycloplegic refraction performed within past 2 months or at the end of the enrollment exam) meets any of the following criteria, then pre-study spectacles are required and must have been worn for at least 1 week prior to enrollment:
* SE anisometropia ≥1.00D
* Astigmatism ≥1.50D in either eye
* SE myopia ≥-1.00D in either eye

Pre-study refractive correction, if worn, must meet the following criteria relative to the cycloplegic refraction performed within past 2 months or at the end of the enrollment exam:

* SE anisometropia must be corrected within <1.00D of the SE anisometropic difference
* Astigmatism must be corrected within <1.00D of full magnitude; axis must be within 10 degrees.
* The SE of the spectacles must not meet the definition of substantial overminus (see exclusion criteria below)
* Gestational age ≥ 32 weeks
* Birth weight > 1500 grams
* Parent understands the protocol and is willing to accept randomization to overminus spectacles or non-overminus spectacles
* Parent has home phone (or access to phone) and is willing to be contacted by Jaeb Center staff and Investigator's site staff
* Relocation outside of area of an active PEDIG site within next 18 months is not anticipated

Exclusion Criteria:

* Treatment for IXT or amblyopia (other than refractive correction) within the past 4 weeks, including vision therapy, patching, atropine, or other penalization.
* Current contact lens wear
* Substantial deliberate overminus treatment within the past 6 months, defined as spectacles overminused by more than 1.00D SE than the cycloplegic refractive error (within 2 months or at the end of the enrollment exam)
* Prior strabismus, intraocular, or refractive surgery (including BOTOX injection)
* Abnormality of the cornea, lens, or central retina
* Down syndrome or cerebral palsy
* Severe developmental delay which would interfere with treatment or evaluation (in the opinion of the investigator). Subjects with mild speech delays or reading and/or learning disabilities are not excluded.
* Any disease known to affect accommodation, vergence, and ocular motility such as multiple sclerosis, Graves orbitopathy, dysautonomia, myasthenia gravis, or current use of atropine for amblyopia
* Anti-seizure medications [e.g., carbamazepine (Tegretol, Carbatrol, Epitol, or Equetro), diazepam (Valium or Diastat), clobazam (Frisium or Onfri), clonazepam (Klonopin), lorazepam (Ativan), ethosuximide (Zarontin), felbamate (Felbatol), lacosamide (VIMPAT), gabapentin (Neurontin), oxcarbazepine (Oxtellar XR or Trileptal), phenobarbital, phenytoin (Dilantin or Phenytek), pregabalin (Lyrica), tiagabine (Gabitril), topiramate (Topamax), valproate (Depakote), or zonisamide (Zonegran), vigabatrin (Sabril)]

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 386 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Chen, OD, MS, Study Chair — Marshall B. Ketchum University; S. Ayse Erzurum, MD, Study Chair — Eye Care Associates, Inc.
Locations (61):
- United States (59):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Midwestern University Eye Institute, Glendale, Arizona
  - Arkansas Childrens, Little Rock, Arkansas
  - University Eye Center at Ketchum Health, Anaheim, California
  - Marshall B. Ketchum University, Fullerton, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Saddleback Eye Medical Associates, Mission Viejo, California
  - Stanford University, Palo Alto, California
  - Western University College of Optometry, Pomona, California
  - University of California San Francisco Department of Ophthalmology, San Francisco, California
  - Nova Southeastern University College of Optometry, The Eye Institute, Fort Lauderdale, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - The Emory Eye Center, Atlanta, Georgia
  - St Luke's Hospital, Boise, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Illinois College of Optometry, Chicago, Illinois
  - The Eye Specialists Center, LLC, Chicago Ridge, Illinois
  - Midwestern U Chicago College of Optometry, Downers Grove, Illinois
  - Pediatric Eye Associates, Wilmette, Illinois
  - Indiana University School Of Optometry, Bloomington, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - The Eye Specialist Center, LLC, Munster, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - University of Kentucky Department of Neurology, Lexington, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Wilmer Eye Institute, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Helen DeVos Children's Hospital Pediatric Ophthalmology, Grand Rapids, Michigan
  - Pediatric Ophthalmology, P.C., Grand Rapids, Michigan
  - Children's Eye Care PC, West Bloomfield, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - U of MO St. Louis College of Optometry, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Concord Ophthalmologic Associates, Concord, New Hampshire
  - State University of New York, College of Optometry, New York, New York
  - Duke University Eye Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Ohio State University College of Optometry, Columbus, Ohio
  - Eye Care Associates, Inc., Poland, Ohio
  - Dean A. McGee Eye Institute, University of Oklahoma, Oklahoma City, Oklahoma
  - Pacific University College of Optometry, Portland, Oregon
  - Casey Eye Institute, Portland, Oregon
  - Conestoga Eye, Lancaster, Pennsylvania
  - Salus University/Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - UPMC Children's Eye Center of Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Storm Eye Institute, Charleston, South Carolina
  - Pediatric Eye Specialists, Chattanooga, Tennessee
  - Southern College of Optometry, Memphis, Tennessee
  - Texas Children's Hospital - Dept. Of Ophthalmology, Houston, Texas
  - University of Houston College of Optometry, Houston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - Houston Eye Associates, The Woodlands, Texas
  - Virginia Pediatric Eye Center, Norfolk, Virginia
  - Gundersen Health System, La Crosse, Wisconsin
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - CHU - Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- [Result] Chen AM, Erzurum SA, Chandler DL, Hercinovic A, Melia BM, Bhatt AR, Suh DW, Vricella M, Erickson JW, Miller AM, Marsh JD, Bodack MI, Martinson SR, Titelbaum JR, Gray ME, Holtorf HL, Kong L, Kraker RT, Rahmani B, Shah BK, Holmes JM, Cotter SA; Pediatric Eye Disease Investigator Group. Overminus Lens Therapy for Children 3 to 10 Years of Age With Intermittent Exotropia: A Randomized Clinical Trial. JAMA Ophthalmol. 2021 Apr 1;139(4):464-476. doi: 10.1001/jamaophthalmol.2021.0082. PMID 33662112
- [Derived] Writing Committee for the Pediatric Eye Disease Investigator Group; Pediatric Eye Disease Investigator Group; Chen AM, Erzurum SA, Chandler DL, Hercinovic A, Wu R, Vricella M, Waters AL, Ticho BH, Erickson JW, Han S, McDowell PS, Li Z, Kraker RT, Holmes JM, Cotter SA. Refractive Error Change and Overminus Lens Therapy for Childhood Intermittent Exotropia. JAMA Ophthalmol. 2024 May 1;142(5):417-428. doi: 10.1001/jamaophthalmol.2024.0276. PMID 38536764
- [Derived] Holmes JM, Leske DA, Hercinovic A, Hatt SR, Chandler DL, Li Z, Melia BM, Chen AM, Erzurum SA, Crouch ER, Jenewein EC, Kraker RT, Cotter SA; Pediatric Eye Disease Investigator Group. Rasch-calibrated Intermittent Exotropia Symptom Questionnaire for Children. Optom Vis Sci. 2022 Jun 1;99(6):513-520. doi: 10.1097/OPX.0000000000001901. Epub 2022 Apr 12. PMID 35412528
- See also: PEDIG public website — http://pedig.jaeb.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overminus Treatment | Non-overminus Treatment
Started | 196 | 190
6 mo Follow Up Visit | 188 | 171
12 mo Follow Up Visit | 189 | 169
15 mo Follow Up Visit | 180 | 153
Completed | 176 | 155
Not Completed | 20 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Overminus Treatment | Non-overminus Treatment | Total
Number analyzed (Participants) | 196 | 190 | 386
Age, Customized [Count of Participants; unit: Participants]
  3 to <7 years | 123 | 120 | 243
  7 to <11 years | 73 | 70 | 143
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 114 | 226
  Male | 84 | 76 | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 6 | 10 | 16
  Race/Ethnicity: Black/African American | 34 | 28 | 62
  Race/Ethnicity: Hispanic | 31 | 40 | 71
  Race/Ethnicity: White | 113 | 91 | 204
  Race/Ethnicity: Other | 12 | 21 | 33
Refractive Error [Count of Participants; unit: Participants]
  >0.50 Diopters | 58 | 59 | 117
  >-0.75 to 0.50 Diopters | 101 | 96 | 197
  -0.75 to >-3.00 Diopters | 29 | 32 | 61
  <=-3.00 Diopters | 8 | 3 | 11
Prior Non Surgical Treatment of IXT [Count of Participants; unit: Participants]
  None | 126 | 137 | 263
  Patching only | 53 | 33 | 86
  Vision therapy only | 10 | 11 | 21
  Patching plus other | 4 | 6 | 10
  Other | 3 | 3 | 6
Randot Preschool Stereoacuity test score at near [Count of Participants; unit: Participants] — Population: Eight participants in the overminus group (5%) and 7 in the nonoverminus group (7%) did not understand test instructions to complete the stereotest; therefore, their stereoacuity at baseline was missing.
  Participants
    number analyzed (Participants) | 188 | 183 | 371
    40-100 arcseconds | 120 | 112 | 232
    200-800 arcseconds | 52 | 55 | 107
    Nil | 16 | 16 | 32
Mean distance visual acuity [Count of Participants; unit: Participants]
  20/12 to 20/20 | 115 | 112 | 227
  20/25 to 20/32 | 70 | 69 | 139
  20/40 to 20/50 | 11 | 9 | 20
IOD of distance visual acuity [Count of Participants; unit: Participants]
  0 lines | 130 | 115 | 245
  0.1 lines | 57 | 61 | 118
  0.2 lines | 9 | 14 | 23
Spectacle wear [Count of Participants; unit: Participants]
  Does not wear spectacles | 140 | 142 | 282
  Wearing spectacles for at least 1 week | 56 | 48 | 104
Exotropia Control at Distance [Count of Participants; unit: Participants] — Control of the exodeviation was measured at distance and near using the IXT Office Control Score, (Mohney, 2006) which ranges from 0 (phoria) to 5 (constant exotropia). Control levels 3-5 were assigned based on the duration of manifest exotropia during a 30-second period before any dissociation. If no exotropia was observed, control levels 0-2 were assigned based on the longest time to reestablishing fusion after 3 consecutive 10-second periods of dissociation. Control was measured at the beginning, middle, and end (3 tests) of a 20- to 40-minute office examination, and the mean was used.
  Participants
    0 to <1 points | NA — Eligibility criteria required distance control at baseline to be at least 2 points | NA — Eligibility criteria required distance control at baseline to be at least 2 points | NA — Total not calculated because data are not available (NA) in one or more arms.
    1 to <2 points | NA — Eligibility criteria required distance control at baseline to be at least 2 points | NA — Eligibility criteria required distance control at baseline to be at least 2 points | NA — Total not calculated because data are not available (NA) in one or more arms.
    2 to <3 points | 84 | 78 | 162
    3 to <4 points | 56 | 52 | 108
    4 to 5 points | 56 | 60 | 116
Exotropia Control at near [Count of Participants; unit: Participants] — Control of the exodeviation was measured at distance and near using the IXT Office Control Score, (Mohney, 2006) which ranges from 0 (phoria) to 5 (constant exotropia). Control levels 3-5 were assigned based on the duration of manifest exotropia during a 30-second period before any dissociation. If no exotropia was observed, control levels 0-2 were assigned based on the longest time to reestablishing fusion after 3 consecutive 10-second periods of dissociation. Control was measured at the beginning, middle, and end (3 tests) of a 20- to 40-minute office examination, and the mean was used.
  Participants
    0 to <1 points | 37 | 46 | 83
    1 to <2 points | 80 | 65 | 145
    2 to <3 points | 39 | 44 | 83
    3 to <4 points | 31 | 27 | 58
    4 to 5 points | 9 | 8 | 17
PACT exodeviation at distance [Count of Participants; unit: Participants] — Δ= prism dipoters
  Participants
    No exodeviation (orthophoria) | NA — PACT at distance was required to be at least 15Δ for eligibility. | NA — PACT at distance was required to be at least 15Δ for eligibility. | NA — Total not calculated because data are not available (NA) in one or more arms.
    1-9 Δ | NA — PACT at distance was required to be at least 15Δ for eligibility. | NA — PACT at distance was required to be at least 15Δ for eligibility. | NA — Total not calculated because data are not available (NA) in one or more arms.
    10-15 Δ | 5 | 6 | 11
    16-18 Δ | 42 | 22 | 64
    19-25 Δ | 86 | 91 | 177
    30-35 Δ | 54 | 50 | 104
    40-45 Δ | 9 | 19 | 28
    >= 50 Δ | 0 | 2 | 2
    Esodeviation | NA — PACT at distance was required to be at least 15Δ for eligibility. | NA — PACT at distance was required to be at least 15Δ for eligibility. | NA — Total not calculated because data are not available (NA) in one or more arms.
PACT Exodeviation at near [Count of Participants; unit: Participants] — Δ= prism diopters
  Participants
    No Exodeviation (orthophoria) | 2 | 3 | 5
    1-9 Δ | 27 | 24 | 51
    10-15 Δ | 45 | 45 | 90
    16-18 Δ | 36 | 29 | 65
    19-25 Δ | 57 | 59 | 116
    30-35 Δ | 24 | 21 | 45
    40-45 Δ | 4 | 8 | 12
    >= 50 Δ | 1 | 0 | 1
    Esodeviation | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance Control at 12-Months (On-Treatment Visit)
Description: A comparison of mean control of the distance exodeviation (average of 3 measurements over the exam) between the 2.50 diopters (D) overminus group and the non-overminus group (spectacles without overminus or no spectacles) at 12 months. The Office Control Score provides a rating of exodeviation control on a 0 to 5 scale, in subjects with intermittent exotropia. Scores 3 to 5 reflect the proportion of time a spontaneous manifest exotropia is present during 30 seconds of observation (<50% score 3; >50% score 4; 100% score 5). If no spontaneous manifest exotropia is observed, scores 0 to 2 reflect the longest time to regain fusion after three, 10-second dissociations (>5 seconds score 2; 1-5 seconds score 1; <1 second score 0).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
points | 1.8 (1.3) | 2.8 (1.5)

2. Primary Outcome: Mean Distance Control at 18-Months (Off-Treatment Visit)
Description: A comparison of mean control of the distance exodeviation (average of 3 measurements over the exam) between the 2.50D overminus group and the non-overminus group (spectacles without overminus or no spectacles) at 18 months (after treatment discontinuation). The Office Control Score provides a rating of exodeviation control on a 0 to 5 scale, in subjects with intermittent exotropia. Scores 3 to 5 reflect the proportion of time a spontaneous manifest exotropia is present during 30 seconds of observation (<50% score 3; >50% score 4; 100% score 5). If no spontaneous manifest exotropia is observed, scores 0 to 2 reflect the longest time to regain fusion after three, 10-second dissociations (>5 seconds score 2; 1-5 seconds score 1; <1 second score 0).
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
points | 2.4 (1.5) | 2.7 (1.6)

3. Secondary Outcome: Number of Participants With No Spontaneous Tropia
Description: The number of subjects with no spontaneous tropia at 12 months and at 18 months will be compared between treatment groups.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
Participants | 115 | 62

4. Secondary Outcome: No Spontaneous Tropia
Description: The proportion of subjects with no spontaneous tropia at 12 months and at 18 months will be compared between treatment groups.
Time Frame: At 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
Participants | 85 | 60

5. Secondary Outcome: Change in Distance Control
Description: The proportion of subjects with ≥1 point improvement in distance control between baseline and 12 months will be compared between treatment groups. The proportion of subjects with ≥2 points improvement in distance control will be similarly compared between treatment groups. The Office Control Score provides a rating of exodeviation control on a 0 to 5 scale, in subjects with intermittent exotropia. Scores 3 to 5 reflect the proportion of time a spontaneous manifest exotropia is present during 30 seconds of observation (<50% score 3; >50% score 4; 100% score 5). If no spontaneous manifest exotropia is observed, scores 0 to 2 reflect the longest time to regain fusion after three, 10-second dissociations (>5 seconds score 2; 1-5 seconds score 1; <1 second score 0).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
Participants
  >1 Point | 116 | 71
  >2 Points | 65 | 24
Statistical Analysis 1: Comparison: Overminus Treatment; >1 point analysis; Test type: Other; Risk Difference (RD) = 19, 95% CI 2-sided [7 to 29]
Statistical Analysis 2: Comparison: Overminus Treatment; Test type: Other — >2 points analysis; Risk Difference (RD) = 20, 95% CI 2-sided [10 to 28]

6. Secondary Outcome: Change in Distance Control
Description: The proportion of subjects with ≥1 point improvement in distance control between baseline and 18 months will be compared between treatment groups. The proportion of subjects with ≥2 points improvement in distance control will be similarly compared between treatment groups. The Office Control Score provides a rating of exodeviation control on a 0 to 5 scale, in subjects with intermittent exotropia. Scores 3 to 5 reflect the proportion of time a spontaneous manifest exotropia is present during 30 seconds of observation (<50% score 3; >50% score 4; 100% score 5). If no spontaneous manifest exotropia is observed, scores 0 to 2 reflect the longest time to regain fusion after three, 10-second dissociations (>5 seconds score 2; 1-5 seconds score 1; <1 second score 0).
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
Participants
  >1 Point | 86 | 68
  >2 Points | 48 | 30
Statistical Analysis 1: Comparison: Overminus Treatment; Test type: Other — >1 analysis; Risk Difference (RD) = 4, 95% CI 2-sided [-7 to 15]
Statistical Analysis 2: Comparison: Overminus Treatment; Test type: Other — >2 analysis; Risk Difference (RD) = 8, 95% CI 2-sided [-2 to 17]

7. Secondary Outcome: Deterioration as Assessed by Motor Alignment and Stereoacuity at Near (12 Months)
Description: The cumulative proportion of subjects who meet deterioration criteria by the time point will be estimated for each treatment group.
  Participants who meet either of the following at any visit by a specific timepoint (e.g., 12 months, 18 months) will be considered to have met deterioration criteria by that timepoint.
  * Motor deterioration: Control of the exodeviation measures 5 (constant exotropia) on all three assessments at distance and near. The exodeviation does not need to be constant throughout the entire exam provided that it is constant during all three assessments of control.
  * Stereoacuity deterioration: Drop in near stereoacuity of at least 2 octaves from enrollment stereoacuity, or to nil, confirmed by a retest by a Masked Examiner on a subsequent day.
  Note: participants with nil stereoacuity at enrollment will not be able to deteriorate with respect to a drop in near stereoacuity.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
Participants | 5 | 7

8. Secondary Outcome: Deterioration as Assessed by Motor Alignment and Stereoacuity at Near (18 Months)
Description: as for outcome 7
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
Participants | 6 | 16

9. Secondary Outcome: Near Control (12 Months)
Description: Mean control of the near exodeviation (average of 3 measurements over the exam). The Office Control Score provides a rating of exodeviation control on a 0 to 5 scale, in subjects with intermittent exotropia. Scores 3 to 5 reflect the proportion of time a spontaneous manifest exotropia is present during 30 seconds of observation (<50% score 3; >50% score 4; 100% score 5). If no spontaneous manifest exotropia is observed, scores 0 to 2 reflect the longest time to regain fusion after three, 10-second dissociations (>5 seconds score 2; 1-5 seconds score 1; <1 second score 0).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
Participants
  0 to <1 points | 96 | 64
  1 to <2 points | 59 | 55
  2 to <3 points | 21 | 13
  3 to <4 points | 9 | 17
  4 to 5 points | 4 | 20

10. Secondary Outcome: Near Control (18 Months)
Description: as for outcome 9
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
Participants
  0 to <1 points | 72 | 59
  1 to <2 points | 60 | 46
  2 to <3 points | 16 | 18
  3 to <4 points | 15 | 16
  4 to 5 points | 13 | 16

11. Secondary Outcome: Change in Near Control (12 Months)
Description: For each timepoint, the change in near control since baseline will be reported. The Office Control Score provides a rating of exodeviation control on a 0 to 5 scale, in subjects with intermittent exotropia. Scores 3 to 5 reflect the proportion of time a spontaneous manifest exotropia is present during 30 seconds of observation (<50% score 3; >50% score 4; 100% score 5). If no spontaneous manifest exotropia is observed, scores 0 to 2 reflect the longest time to regain fusion after three, 10-second dissociations (>5 seconds score 2; 1-5 seconds score 1; <1 second score 0).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
points | 0.7 (1.3) | 0.1 (1.4)

12. Secondary Outcome: Change in Near Control (18 Months)
Description: as for outcome 11
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
points | 0.4 (1.4) | 0.1 (1.5)

13. Secondary Outcome: Angle Magnitude (12 Months)
Description: The magnitude of the deviation by Prism Alternate Cover Test (PACT) will be compared between treatment groups.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Prism Diopters
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
Prism Diopters | 20.0 (9.0) | 25.0 (8.0)

14. Secondary Outcome: Angle Magnitude (18 Months)
Description: The magnitude of the deviation by Prism Alternate Cover Test (PACT) will be compared between treatment groups.
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: Prism Diopters
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
Prism Diopters | 23.0 (9.0) | 24.0 (11.0)

15. Secondary Outcome: Stereoacuity at 12 Months
Description: A comparison of near stereoacuity will be assessed using the Randot Preschool stereotest at near (performed at 40 cm) between treatment groups.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: arcseconds
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
arcseconds | 2.0 (0.4) | 2.0 (0.4)

16. Secondary Outcome: Stereoacuity at 18 Months
Description: as for outcome 15
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: arcseconds
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
arcseconds | 1.9 (0.4) | 1.9 (0.4)

17. Secondary Outcome: Compliance With Spectacle Wear (12 Months)
Description: Compliance with spectacle wear will be assessed at the 12-month and 18-month outcome exam. Parents will give an estimate of the proportion of the time their children wore their spectacles. Proportion of time worn will be described as excellent (76% to 100%), good (51% to 75%), fair (26% to 50%), or poor (≤ 25%). The distribution of compliance will be assessed for each treatment group at the outcome exam.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
Participants
  Excellent (76-100%) | 143 | 128
  Good (51-75%) | 26 | 28
  Fair (26-50%) | 10 | 8
  Poor (1-25%) | 6 | 2
  Prescribed not wearing (0%) | 3 | 2
  Discontinued | 1 | 1

18. Secondary Outcome: Compliance With Spectacle Wear (18 Months)
Description: as for outcome 17
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
Participants
  Excellent (76-100%) | 128 | 120
  Good (51-75%) | 23 | 14
  Fair (26-50%) | 8 | 13
  Poor (1-25%) | 9 | 5
  Prescribed not wearing (0%) | 5 | 1
  Discontinued | 3 | 2

19. Secondary Outcome: Parent Symptom Survey [12 Months]
Description: A brief survey of symptoms that may be associated with overminus such as headaches, eye strain, and problems with spectacle wear will be administered to the parents of the subjects. Parents are asked to respond to the survey questions based on their observations of their child in the past 2 weeks. Response options are based on frequency of observations; never, rarely, sometimes, often, always, and not applicable.
Time Frame: At 12 months
Population: When number analyzed differs from full population size, it indicates that those children were not wearing spectacles, and therefore could not answer the spectacle related questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 189 | 169
Participants
  Did your child have headaches?: Missing | 1 | 1
  Did your child have headaches?: Never | 74 | 71
  Did your child have headaches?: Almost never | 58 | 64
  Did your child have headaches?: Sometimes | 46 | 32
  Did your child have headaches?: Often | 7 | 1
  Did your child have headaches?: Almost Always | 3 | 0
  Did your child have eyestrain?: Missing | 1 | 1
  Did your child have eyestrain?: Never | 75 | 56
  Did your child have eyestrain?: Almost never | 43 | 56
  Did your child have eyestrain?: Sometimes | 60 | 50
  Did your child have eyestrain?: Often | 9 | 6
  Did your child have eyestrain?: Almost Always | 1 | 0
  Did your child avoid reading?: Missing | 1 | 1
  Did your child avoid reading?: Never | 112 | 100
  Did your child avoid reading?: Almost never | 46 | 43
  Did your child avoid reading?: Sometimes | 21 | 18
  Did your child avoid reading?: Often | 7 | 5
  Did your child avoid reading?: Almost Always | 2 | 2
  Did your child have blurry vision?: Missing | 1 | 1
  Did your child have blurry vision?: Never | 106 | 105
  Did your child have blurry vision?: Almost never | 41 | 36
  Did your child have blurry vision?: Sometimes | 34 | 26
  Did your child have blurry vision?: Often | 5 | 1
  Did your child have blurry vision?: Almost Always | 2 | 0
  Did your child look over their spectacles?: number analyzed (Participants) | 185 | 167
  Did your child look over their spectacles?: Missing | 1 | 1
  Did your child look over their spectacles?: Never | 66 | 53
  Did your child look over their spectacles?: Almost never | 37 | 40
  Did your child look over their spectacles?: Sometimes | 45 | 52
  Did your child look over their spectacles?: Often | 25 | 17
  Did your child look over their spectacles?: Almost Always | 11 | 4
  Did your child take their spectacles off?: number analyzed (Participants) | 185 | 168
  Did your child take their spectacles off?: Missing | 1 | 1
  Did your child take their spectacles off?: Never | 38 | 32
  Did your child take their spectacles off?: Almost never | 45 | 51
  Did your child take their spectacles off?: Sometimes | 63 | 66
  Did your child take their spectacles off?: Often | 28 | 16
  Did your child take their spectacles off?: Almost Always | 10 | 2
  Did your child complain about hurt ears/nose?: number analyzed (Participants) | 186 | 168
  Did your child complain about hurt ears/nose?: Missing | 1 | 1
  Did your child complain about hurt ears/nose?: Never | 112 | 96
  Did your child complain about hurt ears/nose?: Almost never | 43 | 47
  Did your child complain about hurt ears/nose?: Sometimes | 18 | 22
  Did your child complain about hurt ears/nose?: Often | 10 | 2
  Did your child complain about hurt ears/nose?: Almost Always | 2 | 0

20. Secondary Outcome: Parent Symptom Survey [18 Months]
Description: as for outcome 19
Time Frame: At 18 months
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Overminus Treatment | Non-overminus Treatment
Number analyzed (Participants) | 176 | 155
Participants
  Did your child have headaches?: Missing | 0 | 1
  Did your child have headaches?: Never | 76 | 63
  Did your child have headaches?: Almost never | 49 | 55
  Did your child have headaches?: Sometimes | 46 | 31
  Did your child have headaches?: Often | 4 | 3
  Did your child have headaches?: Almost always | 1 | 2
  Did your child have eyestrain?: Missing | 0 | 1
  Did your child have eyestrain?: Never | 66 | 49
  Did your child have eyestrain?: Almost never | 52 | 50
  Did your child have eyestrain?: Sometimes | 53 | 49
  Did your child have eyestrain?: Often | 3 | 6
  Did your child have eyestrain?: Almost always | 2 | 0
  Did your child avoid reading?: Missing | 0 | 1
  Did your child avoid reading?: Never | 102 | 94
  Did your child avoid reading?: Almost never | 44 | 41
  Did your child avoid reading?: Sometimes | 24 | 14
  Did your child avoid reading?: Often | 4 | 4
  Did your child avoid reading?: Almost always | 2 | 1
  Did your child have blurry vision?: Missing | 0 | 1
  Did your child have blurry vision?: Never | 99 | 92
  Did your child have blurry vision?: Almost never | 46 | 37
  Did your child have blurry vision?: Sometimes | 29 | 23
  Did your child have blurry vision?: Often | 1 | 1
  Did your child have blurry vision?: Almost always | 1 | 1
  Did your child look over their spectacles?: number analyzed (Participants) | 173 | 151
  Did your child look over their spectacles?: Missing | 0 | 1
  Did your child look over their spectacles?: Never | 54 | 55
  Did your child look over their spectacles?: Almost never | 46 | 33
  Did your child look over their spectacles?: Sometimes | 47 | 48
  Did your child look over their spectacles?: Often | 18 | 9
  Did your child look over their spectacles?: Almost always | 8 | 5
  Did your child take their spectacles off?: number analyzed (Participants) | 172 | 152
  Did your child take their spectacles off?: Missing | 0 | 1
  Did your child take their spectacles off?: Never | 38 | 32
  Did your child take their spectacles off?: Almost never | 36 | 43
  Did your child take their spectacles off?: Sometimes | 69 | 55
  Did your child take their spectacles off?: Often | 22 | 13
  Did your child take their spectacles off?: Almost always | 7 | 8
  Did your child complain about hurt ears/nose?: number analyzed (Participants) | 174 | 152
  Did your child complain about hurt ears/nose?: Missing | 0 | 1
  Did your child complain about hurt ears/nose?: Never | 109 | 96
  Did your child complain about hurt ears/nose?: Almost never | 41 | 36
  Did your child complain about hurt ears/nose?: Sometimes | 18 | 14
  Did your child complain about hurt ears/nose?: Often | 2 | 4
  Did your child complain about hurt ears/nose?: Almost always | 4 | 1

ADVERSE EVENTS:
Time Frame: 18 months
Description: Although no adverse events are anticipated as a result of overminus therapy or non-overminus spectacle wear, any new cases of amblyopia, constant esotropia, or constant exotropia at distance and near will be reported. No surgical procedures are part of the protocol and no treatments are being prescribed that are not part of usual care. Investigators will abide by local IRB reporting requirements.
Arm/Group | Overminus Treatment | Non-overminus Treatment
All-Cause Mortality (participants affected / at risk) | 0/196 | 0/190
Serious Adverse Events (participants affected / at risk) | 0/196 | 0/190
Other Adverse Events (participants affected / at risk) | 47/196 | 15/190
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overminus Treatment (N=196) | Non-overminus Treatment (N=190)
Development of Esotropia (Eye disorders) | 4 (4) | 4 (4)
>1 Diopter of Myopic Shift (Eye disorders) | 33 (33) | 2 (2) — DSMC found more participants experienced the myopia progression in the overminus group than the non-overminus group. DSMC agreed the additional myopia progression is not serious, but recommended that any overminus treatment be stopped.
2 or more line decrease in visual acuity (Eye disorders) | 12 (12) | 10 (10)
Amblyopia treatment prescribed by 12 months (Eye disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02807350/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT02807350/SAP_002.pdf
  • Informed Consent Form (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT02807350/ICF_001.pdf